CLINICAL TRIAL: NCT06876051
Title: The Impact of Prenatal Stress Management Program on Maternal Breastfeeding and Neonatal Neurodevelopmental Parameters
Brief Title: Prenatal Intervention of Maternal Stress - Breastfeeding & Infant Neurodevelopment
Acronym: PRIMAS-BIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: General and Maternity Hospital of Athens Elena Venizelou (Other)
Responsible Party: Principal Investigator, Aikaterini Fotiou, MD, MSc, Pediatrician -Neonatologist, Director of Neonatal Dept/NICU, General and Maternity Hospital "Helena Venizelou", Athens, Greece, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1617031875 / 04-07-17; ID 126/04-09-17 (Other: Scientific Committee, H.Venizelou Hospital, Greece); 1617031875/2017 (Other: NKUA, Medical School)
Record Dates: First submitted 2025-02-09; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Stress; Relaxation; Breastfeeding; Infant Behavior; Prenatal Stress
Keywords: breastfeeding; BDNF; Reelin; pregnancy; relaxation techniques; stress management
MeSH Terms: conditions — Breast Feeding; Infant Behavior | interventions — Autogenic Training; Imagery, Psychotherapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Primipara Pregnant women are randomly assigned to one of three groups: (1) an intervention group receiving relaxation techniques combined with breastfeeding education, (2) an active control group receiving only breastfeeding education, and (3) a control group receiving standard maternity care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Behavioral: Relaxation & Breastfeeding Education (Experimental): Participants in the intervention group (primiparous pregnant women) receive:
  1. Training in relaxation techniques, including guided breathing exercises, progressive muscle relaxation, and visualization methods.
  2. Breastfeeding education, covering topics such as proper latching, milk production, and infant feeding schedules.
  The intervention consists of 8-10 structured sessions, beginning in the second trimester (gestational weeks 15-20) and continuing until the 36th week of gestation. Sessions are conducted in a structured format by trained professionals.
  Interventions: Behavioral: Relaxation & Breastfeeding Education
- Behavioral : Breastfeeding Education Alone (Active Comparator): Participants in the Active Comparator group receive 8-10 individual lessons covering: Pregnancy education, Breastfeeding techniques and best practices, Childbirth preparation, Newborn care essentials, Understanding infant cues and responses.
  These sessions are delivered in a structured format by trained professionals. No relaxation techniques are included in this intervention.
  Interventions: Behavioral: Active comparator
- Standard Maternity Care (Control Group) (Other): Participants in the control group receive only the standard maternity care provided by health services during pregnancy.
  The maternity hospital is designated as a Baby-Friendly Hospital and follows its established guidelines and principles.
  Standard care includes routine prenatal check-ups and general health services. The hospital also offers psycho-prophylactic preparation for normal childbirth and one breastfeeding course, both led by midwife trainers.
  No additional intervention, such as relaxation techniques or structured breastfeeding education, is provided to this group.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Relaxation & Breastfeeding Education — Pregnant women in this group will be trained in 10 individual interactive sessions, focusing on relaxation techniques and breastfeeding including:
  1. Diaphragmatic breathing
  2. Progressive muscle relaxation (PMR) - tailored for pregnant women.
  3. Guided imagery
  4. the analysis of the concept of stress and stress management strategies for pregnancy including Cognitive-behavioral approach (CBT principles)
  5. Mindfulness-based pregnancy adaptation including positive thinking and wellbeing during pregnancy .
  6. Pregnancy stages.
  7. Benefits of breastfeeding.
  8. Breastfeeding guide and practical applications.
  9. Labor stages and childbirth preparation.
  10. Newborn and infant needs at home Every relaxation technique training will last 20 minutes practice in every session Additionally pregnant women will be practiced at least 3 times weekly during pregnancy
  Other Names: Prenatal relaxation techniques; prenatal stress management; prenatal educational breastfeeding programme; diaphragmatic breathing; progressive Muscle Relaxation; Guided Imagery; positive thinking
  Arms: Behavioral: Relaxation & Breastfeeding Education
Behavioral: Active comparator — Participants in this group will receive only interactive online education, focusing exclusively on breastfeeding and newborn care. The Programme included ten remote sessions:
  1. Pregnancy stages.
  2. Benefits of breastfeeding.
  3. Skin-to-skin contact and rooming-in during the first days.
  4. The role of breastfeeding in maternal emotional well-being.
  5. Breastfeeding guide and practical applications.
  6. Maternal nutrition during breastfeeding.
  7. Common breastfeeding challenges.
  8. The father's role in breastfeeding support.
  9. Labor stages and childbirth preparation
  10. Newborn and infant needs at home.
  Other Names: prenatal Breastfeeding Education; Infant cues on breastfeeding; breastmilk benefits; breastfeeding guide
  Arms: Behavioral : Breastfeeding Education Alone
Other: control group — This group will received only standard prenatal and postnatal care at a Baby-Friendly Hospital, which adheres to WHO and UNICEF guidelines for breastfeeding support. They did not participate in additional structured educational programs or relaxation training.
  Other Names: Routine Maternity Care; Baby Friendly Hospital Initiative
  Arms: Standard Maternity Care (Control Group)

SUMMARY:
The goal of this clinical trial is to determine whether antenatal maternal stress management using relaxation techniques improves breastfeeding effectiveness and neonatal neurodevelopmental outcomes. It is hypothesized that reducing maternal stress during pregnancy will enhance the initiation and continuation of exclusive breastfeeding until six months postpartum.

The management of antenatal maternal stress is expected to be reflected in both the newborn's behavior and proteins associated with neurodevelopment, such as Brain-Derived Neurotrophic Factor (BDNF) and Reelin.

The main research questions of this study include the following:

1. Does stress management in pregnant women using relaxation techniques increase the likelihood of exclusive breastfeeding at one and six months postpartum?
2. Does it impact neonatal and infant growth and behavior?
3. Does it alter neurotrophin levels in the fetus? This trial will provide insight into the potential benefits of prenatal stress reduction for both maternal and infant health outcomes.
4. "If prenatal stress management leads to changes in neurotrophins in the fetus, could these changes be linked to the success and duration of breastfeeding, as well as the infant's growth and behavior?

DETAILED DESCRIPTION:
METHODOLOGY Researchers will compare three groups of pregnant women who will receive three different types of information during pregnancy.

* The first group, or intervention group (IG), will be trained in 8-10 structured individual sessions of relaxation techniques that they will apply throughout the pregnancy, along with structured information about breastfeeding.
* The second group, or Active Control group (ACG), will receive 8 individual structured educational courses about breastfeeding, childbirth and the needs of the newborn, and
* The third group, or Control Group (CG), will receive a standard use information provided by the hospital midwife stuff about childbirth and breastfeeding in 3-4 group meetings .

Participants will be primipara pregnant women native speaking of the Greek language and they will be included in the study after randomization based on the electronic system random.org , between the 15th and 20th week of gestation They will be studied in 4 time periods (phases) .

* The first phase, will be prenatally at the beginning of the study between 15th -20th week of gestation,
* the second phase, will be prenatally at the end of the study between the 34th and 36th week of gestation,
* the third phase, will be in the first month after childbirth and
* the fourth phase, will be in the 6th month of their baby's life. The study as well, will include the newborns of the participants in the third and fourth phase of the study, corresponding them to the group of their mothers.

Comparisons will be in each group and between the groups investigating the alteration of stress, anxiety and depression during the four time periods pre and postnatally . Concurrently the change in the belief of successful breastfeeding during the two first periods of time (phase 1 and 2 ) , prenatally, will be compared with the real outcome at the phase 3 and 4.

For each participant, the following data will be recorded:

Phases 1 and 2:

1. Demographic data
2. Pregnancy stress, assessed using the Prenatal Experience Brief Scale
3. Pregnancy anxiety, assessed using the Pregnancy Anxiety Questionnaire
4. Prenatal breastfeeding self-efficacy, assessed using the Prenatal e. Breastfeeding Self-Efficacy Scale

Phases 1, 2, 3, and 4:

1. Perceived stress, assessed using the Perceived Stress Scale-14 (PSS-14)
2. Postpartum depression, assessed using the Edinburgh Postpartum Depression Scale (EPDS)
3. Anxiety, assessed using the Spielberger State-Trait Anxiety Inventory (STAI)

Phases 3 and 4:

1. Breastfeeding self-efficacy, assessed using the Breastfeeding Self-Efficacy Scale
2. Breastfeeding-related questions from the Pregnancy Risk Assessment Monitoring System (PRAMS) of the CDC

Phase 4 only :

1. Maternal attachment, assessed using the Maternal Attachment Scale
2. Infant behavior, assessed using the Infant Behavior Questionnaire

For each newborn, the following data will be recorded:

1. Anthropometric measurements at birth (3rd phase) and at six months of age (4th phase).
2. Neonatal behavior, assessed between the 4th and 7th day of life (3rd phase) using the Neonatal Behavioral Assessment Scale (NBAS). The evaluation will be conducted by a healthcare professional trained and familiar with the use of this specific behavioral assessment tool.
3. Developmental milestones at six months of age (4th phase).
4. Infant behavior assessment at six months of age (4th phase), conducted using the Infant Behavior Questionnaire, which will be completed by the parents based on their own observations and assessment

Biological Markers Collection and Analysis

The collection of biological markers is structured according to the study phase:

* In phases 1 and 2, salivary cortisol will be measured in pregnant participants. Participants will be asked to collect saliva using Salivettes (Sarstedt), following specific instructions provided by the manufacturer.
* In phases 1 and 3, maternal serum neurotrophins (BDNF and Reelin) will be analyzed. Additionally, in phase 3, umbilical cord serum neurotrophins will be measured.

Saliva Collection and Analysis

Saliva collection will be conducted at four time points throughout the day to assess the circadian rhythm of each pregnant participant:

* Morning, immediately upon awakening
* 30 minutes after awakening
* Afternoon, before lunch (around 3:00 PM)
* Night, before bedtime (around 12:00 AM) Pregnant participants will store the collected samples in the refrigerator until they bring them to the laboratory the following day. At the laboratory, the samples will undergo centrifugation followed by measurement using Chromatography/Mass Spectrometry.. The saliva samples will be centrifuged for 2 minutes at 1,000 × g, following the manufacturer's instructions.

Neurotrophin Measurement (BDNF & Reelin) - Phases 1 and 3

The measurement of BDNF and Reelin neurotrophins will be performed on serum blood samples collected at three time points:

1. Phase 1: At the start of the intervention (between 15-20 weeks of gestation) - maternal blood serum.
2. Phase 3: Before delivery (at hospital admission, marking the end of the prenatal intervention) - maternal blood serum.
3. Phase 3: During delivery - umbilical cord serum only. All blood samples will undergo centrifugation at 3500 rpm for 5-6 minutes. The separated serum will then be transferred into Eppendorf tubes and stored at -80°C until further analysis. Neurotrophin levels (BDNF & Reelin) will be measured using the ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women
* 14-20 weeks of Gestational Age
* Intention to give birth at the specific maternity hospital
* Greek women or foreigners who know the Greek language very well
* Place of residence: Greece

Exclusion Criteria:

* Use of benzodiazepines, major neuroleptics, or psychostimulant medications.
* Pregnant women diagnosed with incurable physical or mental diseases.
* Pregnant women carrying fetuses or newborns with major congenital anomalies or criteria for perinatal asphyxia.
* Pregnant women with stillbirths or newborns who do not survive.
* All mothers and their newborns born before 34 weeks of gestation or requiring hospitalization in the Neonatal Intensive Care Unit (NICU) for more than 7 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes only primiparous pregnant women from the beginning of the second trimester until the end of the 36th gestational week.
Enrollment: 162 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Prenatal Breastfeeding Self-Efficacy Across Study Groups | 1) between 15 - 20 week of gestation and 2) between 35-38 weeks gestation before child birth
  This outcome will assess maternal confidence in breastfeeding and actual breastfeeding before childbirth using the Prenatal Breastfeeding Self-Efficacy Scale (PBSES), a validated tool that measures prenatal maternal perceived ability to breastfeed successfully. The PBSES consists of 20 items rated on a 5-point Likert scale, with a SUM score ranging from 20 (minimum) to 100 (maximum). Scores will be recorded without a cutoff point, with higher scores indicating greater prenatal maternal confidence in breastfeeding. Comparisons will be conducted among the three study groups to evaluate differences in PBSES scores based on the intervention received.
  Statistical analysis will include the comparisons across study groups using ANOVA or non-parametric equivalents. Regression models to explore potential predictors of higher or lower prenatal self-efficacy.
Breastfeeding Self-Efficacy across the study groups and the time frames | At 1 and 6 months postpartum
  Maternal breastfeeding self-efficacy will be assessed using the Breastfeeding Self-Efficacy Scale (BSES), a validated questionnaire measuring maternal confidence in breastfeeding. The BSES consists of 14 items, each rated on a 5-point scale (1 = Strongly Disagree, 5 = Strongly Agree). The final score is calculated as the sum of all item scores, with higher scores indicating greater breastfeeding self-efficacy. Minimum Value is 14 (lowest BSES score) and Maximum Value is70 (highest BSES score) Comparative analyses will be conducted across the three study groups to evaluate differences in self-efficacy levels.
Breastfeeding Outcomes Across Study Groups | at 1 and 6 Months Postpartum
  Breastfeeding outcomes will be derived from responses to selected PRAMS questions, which indirectly indicate exclusivity. Breastfeeding success will be numerically categorized (1 = Exclusive breastfeeding, 2 = Any breastfeeding, 3 = No breastfeeding) to allow for statistical comparison with Breastfeeding Self-Efficacy Scale (BSES) scores. The analysis will examine whether higher BSES scores are associated with exclusive or any breastfeeding.
Neurotrophin Levels as Neurodevelopmental Parameters in Maternal Serum and Umbilical Cord Blood across the study groups | In Maternal serum: 1) between the 15th -20th weeks of gestation and 2) at 36-37 weeks of gestation .Additionally Neurotrophins will be measured In Umbilical cord blood: At birth
  The levels of neurotrophins, specifically brain-derived neurotrophic factor (BDNF) and Reelin, will be assessed as neurodevelopmental biomarkers in maternal serum at 15-20 weeks and 36-37 weeks of gestation, and in umbilical cord blood at birth.
  Neurotrophin quantification will be performed using the Enzyme-Linked Immunosorbent Assay (ELISA) method, following standardized protocols.
  Results will be expressed in picograms per milliliter (pg/mL), and comparative analyses will be conducted to evaluate differences across the three study groups and at different time points.
Neonatal Behavioral Assessment Across Study Groups | 4-7 days postpartum
  Neonatal behavior will be assessed using the Neonatal Behavioral Assessment Scale (NBAS), conducted by a personnel trained in administering and scoring the instrumental tool . NBAS contains a large number of individual items scored on a 9-point scale and reflexes scored on a 4-point scale . The evaluated items will be categorized into eight clusters, with scores representing the mean of the item scores within each cluster. The clusters and the number of items per cluster are: 1. Habituation (4 items) , 2. Social -Interactive (7 items) , 3. Motor System (5 items), 4. State Organization(4 items), 5. State Regulation (4 items), 6. Autonomic System (3 items) , 7. Reflexes (18 items), 8. Supplementary Items (7 items)-Additional behavioral observations.
Infant Behavioral Assessment Across Study Groups | IBQ-R SF will be measured at 6 months postpartum
  Infant behavior will be assessed using the Infant Behavior Questionnaire-Revised Short Form (IBQ-R SF), completed by parents. The IBQ-R SF consists of 91 items, each rated on a 7-point Likert scale (1 = Never, 7 = Always). Scores are averaged within each of the 14 behavioral subscales, which are further grouped into three broad temperament dimensions. The final score for each subscale or dimension is calculated as the mean of the corresponding item scores, providing a standardized numerical measurement of infant temperament for comparative analyses across the three study groups.

SECONDARY OUTCOMES:
Correlation Between Maternal age and Breastfeeding success | breastfeeding outcomes : at 1 and 6 month postpartum.
  This outcome measure will assess the correlation between maternal age (in years) and breastfeeding success across the three study groups.
  Breastfeeding success will be categorized as:
  1. = No breastfeeding
  2. = Any breastfeeding
  3. = Exclusive breastfeeding Data will be collected using structured PRAMS-based questions.
  Statistical analysis:
  Pearson's or Spearman's correlation coefficient (r-value) will be used to assess the relationship between maternal age and breastfeeding success.
  Chi-square tests (χ²) will be used for categorical comparisons.
  Multivariate regression analysis will adjust for potential confounders.Unit of Measure:
  Maternal age: Years (continuous variable) Breastfeeding success: Categorical classification (1, 2, 3)
  Higher Scores Mean:
  For maternal age: Not applicable (continuous variable) For breastfeeding success: Higher values (3) indicate better outcomes (exclusive breastfeeding)
Correlation Between Maternal Socioeconomic Status and Breastfeeding success | Household income will be assessed between the 15th and 20th week of gestation, while breastfeeding outcomes will be measured at 1 and 6 months postpartum.
  This outcome measure will assess the correlation between household income and breastfeeding success across the three study groups. Household income will be categorized into six levels based on self-reported data collected between the 15th and 20th week of gestation: 1 = Indigent, 2 = <10,000, 3 = 10,000-20,000, 4 = 20,000-30,000, 5 = 30,000-40,000, and 6 = >40,000. Breastfeeding success will be categorized as 1 = No breastfeeding, 2 = Any breastfeeding, and 3 = Exclusive breastfeeding, based on structured PRAMS-based questions. Statistical analysis will include Spearman's correlation coefficient (r-value) to assess the relationship between household income and breastfeeding success. Chi-square tests (χ²) will be used for categorical comparisons, and multivariate regression analysis for potential confounders. Unit of Measure: Household income will be recorded as an ordinal variable (1-6), and breastfeeding success as a categorical variable (1-3)
correlation of maternal Body Mass Index (BMI) and Breastfeeding success across the three study groups. | BMI assessment: Pre-pregnancy (self-reported) and at delivery (clinically measured) Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Maternal BMI will be calculated as weight (kg) divided by height squared (m²) and recorded at two time points: before pregnancy (self-reported) and at the time of delivery (measured clinically). Maternal BMI: kg/m²
  Breastfeeding success will be assessed using structured PRAMS-based questions, categorizing success as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between maternal BMI and breastfeeding outcomes using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and delivery mode.
Correlation Between Anxiety and Breastfeeding success | STAI assessment: prenatally at 15-20 and 35-38 weeks of gestation . Postnatally, Breastfeeding outcomes assessment: at 1 and 6 months postpartum.
  Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI), a validated self-report questionnaire measuring state and trait anxiety, with each subscale consisting of 20 items rated on a 4-point Likert scale, leading to a SUM score range of 20-80 per subscale.
  Breastfeeding success will be categorized using PRAMS-based structured questions as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between STAI scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and delivery mode.
Correlation Between Pregnancy-Related Anxiety (PRAQ-R2) and Breastfeeding Success across study groups | PRAQ-R2 assessment: Between 15-20 and 35-38 weeks of gestation Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Pregnancy-related anxiety will be assessed using the Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2), a validated self-report questionnaire consisting of 11 items rated on a 5-point Likert scale (1 = Not at all relevant, 5 = Completely relevant), resulting in a SUM score ranging from 11 (lowest anxiety) to 55 (highest anxiety).
  Breastfeeding success will be categorized using PRAMS-based structured questionnaires as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between PRAQ-R2 scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and delivery mode.
Influence of Neonatal Behavior on Breastfeeding Outcomes | NBAS is evaluating between the first 4-7 days of life. Breastfeeding assessment will be at 1 and 6 months postpartum
  This outcome measure examines how neonatal behavior influences breastfeeding success across study groups. Neonatal behavior will be assessed using the Neonatal Behavioral Assessment Scale (NBAS) between the 3rd and 7th day postpartum, evaluating responses to stimuli, alertness, and sucking reflex. Breastfeeding success will be categorized as exclusive, partial, or no breastfeeding, based on structured breastfeeding questionnaires. Additional data will capture early neonatal feeding behaviors, such as skin-to-skin contact, first latch attempts, and initial feeding difficulties. Comparative analyses will assess differences between study groups, while correlation and regression models will explore whether more adaptive neonatal behaviors are associated with higher breastfeeding success rates.
Correlation Between Neurotrophin Levels and Breastfeeding Self-Efficacy across the study groups | Neurotrophin levels: Maternal serum (15-20 and 36-37 weeks gestation), Umbilical cord blood (at birth) Breastfeeding self-efficacy: 1 and 6 months postpartum
  This outcome measure examines the correlation between neurotrophin levels (BDNF, Reelin) and maternal breastfeeding self-efficacy across the three study groups. Neurotrophin levels will be measured in maternal serum and in umbilical cord blood using ELISA (pg/mL). Breastfeeding self-efficacy will be measured using the Breastfeeding Self-Efficacy Scale (BSES) with SUM score (Range: 14-70) Statistical analyses will include Spearman's or Pearson's correlation coefficients, with regression models adjusting for confounders.
Correlation between Prenatal Breastfeeding Self-Efficacy and Breastfeeding Outcomes Across Study Groups | PBSES assessment: 15-20 weeks and 35-38 weeks of gestation Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Maternal breastfeeding self-efficacy will be assessed prenatally using the Prenatal Breastfeeding Self-efficacy Scale (PBSES), consisting of 20 items rated on a 5-point Likert scale (SUM score range: 20-100), to assess maternal confidence in breastfeeding during pregnancy. There are no cut-off points. As the scores get higher, the prenatal breastfeeding self-efficacy increases. Breastfeeding success will be categorized numerically as: 1 = No breastfeeding , 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will examine correlations between prenatal breastfeeding self-efficacy, and breastfeeding success.
  For PBSES: Higher scores indicate greater prenatal breastfeeding For breastfeeding success: Higher values indicate greater breastfeeding success.
Correlation between Postnatal Breastfeeding Self-Efficacy and Breastfeeding Outcomes Across Study Groups | BSES assessment: 1 and 6 months postpartum Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Postnatal breastfeeding self-efficacy will be assessed using the Breastfeeding Self-Efficacy Scale (BSES), a validated questionnaire consisting of 14 items rated on a 5-point Likert scale (SUM score range: 14-70).
  Breastfeeding outcomes will be evaluated using structured PRAMS-based questions, categorizing success as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between postnatal BSES scores and breastfeeding outcomes using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders.
Correlation between Salivary Cortisol levels and Breastfeeding outcomes across the study groups | Salivary cortisol levels at 35-38 week of gestation . Breastfeeding success at 1 month postpartum
  Salivary cortisol will be measured prenatally, using Salivette (Sarstedt) devices and analyzed via Chromatography/Mass Spectrometry (nmol/L).
  Breastfeeding outcomes will be evaluated using structured PRAMS-based questions, categorizing success as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between prenatal maternal cortisol levels and breastfeeding outcomes using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders.
Correlation Between Infant Behavior and Breastfeeding Success across the three study groups | IBQ-R SF assessment: 6 months postpartum Breastfeeding outcomes assessment: 6 months postpartum
  Infant behavior will be assessed at 6 months postpartum using the Infant Behavior Questionnaire-Revised Short Form (IBQ-R SF), a validated parental-report measure of temperament. Breastfeeding success will be categorized as 1 = No breastfeeding, 2 = Partial breastfeeding, 3 = Exclusive breastfeeding, based on structured breastfeeding questionnaires. Unit of Measure: IBQ-R SF score: Mean score per subscale (temperament domains) Breastfeeding success: Categorical classification (1 = No breastfeeding, 2 = Partial breastfeeding, 3 = Exclusive breastfeeding) Statistical analyses will assess correlations between IBQ-R SF scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders.
correlation between newborn hospitalization and breastfeeding success across the study groups | Neonatal hospitalization assessment: At birth Breastfeeding outcomes assessment: 1 and 6 months postpartum
  This outcome measure examines the correlation between neonatal hospitalization (Yes/No) and breastfeeding success across the three study groups. Neonatal hospitalization will be defined as admission to the Neonatal Intensive Care Unit (NICU) or other specialized care units after birth, and recorded as a binary variable (Yes = 1, No = 0).
  Breastfeeding success will be categorized based on structured PRAMS-based questions as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess associations between neonatal hospitalization and breastfeeding success using Chi-square tests (χ²) for categorical comparisons, while logistic regression models will adjust for potential confounders such as gestational age, birth weight, and maternal health factors. For neonatal hospitalization: Not applicable (binary variable) For breastfeeding success: Higher values indicate greater breastfeeding success
Correlation of Breastfeeding difficulties and postpartum breastfeeding support with breastfeeding success across the study groups | Assessment of breastfeeding difficulties and postpartum support: 4 days postpartum Breaffeidng success at 1 and 6 months after birth
  Breastfeeding difficulties will be assessed using 11 PRAMS-based questions, where each item is answered as Yes (2) or No (1), resulting in a SUM score ranging from 11 (minimum difficulties) to 22 (maximum difficulties).
  Postpartum breastfeeding support from maternity hospital staff will be evaluated using 12 PRAMS-based questions, where each item is answered as Yes (2) or No (1), leading to a SUM score ranging from 12 (lowest support) to 24 (highest support).
  Breastfeeding success will be categorized based on PRAMS-based structured questionnaires, as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between breastfeeding difficulties, postpartum support, and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and delivery mode.
Correlation Between Mode of Delivery and Breastfeeding Success across the study groups | Mode of delivery assessment: At birth Breastfeeding outcomes assessment: 1 and 6 months postpartum
  This outcome measure examines the correlation between mode of delivery and breastfeeding success across the three study groups. Mode of delivery will be categorized as follows:
  1 = Cesarean section 2 = Vaginal delivery 3 = Vaginal delivery with induction 4 = Induction attempted for vaginal delivery but resulted in cesarean section 5 = Cesarean section with general anesthesia 6 = Emergency cesarean section Breastfeeding success will be categorized using PRAMS-based structured questionnaires as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between mode of delivery and breastfeeding success using Spearman's or Pearson's correlation coefficients, while logistic regression models will adjust for confounders such as maternal age, socioeconomic status, and gestational age at birth.
  Units of Measure are Mode of delivery: Categorical classification (1-6) Breastfeeding success: Categorical classification (1 - 3)
Correlation Between Postpartum Depression (EPDS) and Breastfeeding Success across the study groups | EPDS assessment: postnatally 1 and 6 months postpartum nad prenatally at 35-38 week of gestation Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Postpartum depression symptoms will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-report questionnaire, where each item is rated on a 4-point Likert scale (0-3), resulting in a SUM score ranging from 0 (no depressive symptoms) to 30 (severe depressive symptoms). Cutoff point will be 10 .
  Breastfeeding success will be categorized using PRAMS-based structured questionnaires as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between EPDS scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and mode of delivery.
Correlation Between Stressful Life Events (Holmes and Rahe Stress Scale) and Breastfeeding Success | Assessment of stressful life events: During pregnancy for the last year . Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Stressful life events will be assessed using the Holmes and Rahe Stress Scale, a validated tool that assigns weighted scores to 43 life events during the last year based on their relative stress impact. The total score is calculated as a SUM score, with higher values indicating greater exposure to stress and increased health risk. Breastfeeding success will be categorized using PRAMS-based structured questionnaires as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding. Statistical analyses will assess correlations between Holmes and Rahe Stress Scale scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal age, socioeconomic status, and mode of delivery.Unit of Measure: Holmes and Rahe Stress Scale score: SUM score (higher values indicate greater exposure to stress) and Breastfeeding success: Categorical classification (1-3)

OTHER OUTCOMES:
Correlation of Mother-child attachment and breastfeeding success | At 6 months postpartum
  Maternal attachment will be assessed using the Maternal Postnatal Attachment Scale (MPAS). The MPAS consists of 19 items, with different item scoring ranging from two-point to five-point scaling. Items are re-coded prior to analysis for equal weighting, with final item scores ranging from 1 to 5. The maximum score is 95, and the theoretical minimum is 19. Lower scores indicate more problematic responses. The MPAS does not have validated cut off points. Higher scores indicate more optimal mother-infant bonding. Breastfeeding success will be categorized as 1 = No breastfeeding, 2 = Partial breastfeeding, 3 = Exclusive breastfeeding, based on structured breastfeeding questions. Statistical analyses will assess correlations between MPAS scores and breastfeeding success using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders.
Correlation of Neonatal and Infant Anthropometric parameters with breastfeeding success across the study groups | Neonatal anthropometric measurements: At birth Infant anthropometric measurements: 1 and 6 months postpartum Breastfeeding outcomes assessment: 1 and 6 months postpartum
  Neonatal anthropometric measurements, including birth weight, body length, and head circumference, will be recorded at birth. Infant anthropometric parameters, including weight, length, and head circumference, will be assessed at 6 months postpartum during routine clinical visit. Units of Measure are for Birth weight & infant weight in kilograms (kg), Body length & head circumference in Centimeters (cm) Breastfeeding success will be categorized as 1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding, based on structured PRAMS-based questions. Statistical analyses will assess correlations between anthropometric parameters and breastfeeding outcomes using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders such as maternal BMI, gestational age, and birth complications.
  Breastfeeding success: Categorical classification (1 = No breastfeeding, 2 = Any breastfeeding, 3 = Exclusive breastfeeding)
Correlation Between prenatal Cortisol Levels and Perceived Stress (PSS-14) | Prenatal cortisol & PSS-14 assessment: 15-20 and 35-38 weeks of gestation. Postnatal PSS-14 assessment: 1 and 6 months postpartum
  This outcome measure examines the correlation between maternal cortisol levels and perceived stress as measured by the Perceived Stress Scale (PSS-14) pre and postnatally across the three study groups and between the time frames. Salivary cortisol will be measured prenatally using Salivette (Sarstedt) devices and analyzed via Chromatography/Mass Spectrometry (nmol/L). PSS-14, is a validated self-report questionnaire that evaluates maternal stress levels on a 5-point Likert scale (from Never = 0 to Very often = 4).Total score of the scale is the sum of all 14 item scores with range 0 (lowest stress) to 56 (highest stress).
  Higher scores indicate greater perceived stress. Statistical analyses will assess correlations between cortisol levels and PSS-14 scores using Pearson's or Spearman's correlation coefficients, while regression models will adjust for potential confounders.
Relationship Between Cortisol Levels and Prenatal Maternal Stress | prenatally : between 15-20 week of gestation and 2) between 35-38 of gestation
  Τhis outcome measure examines the relationship between maternal cortisol levels and prenatal stress as measured by the Pregnancy Experience Scale Brief (PES-brief) across the three study groups. Salivary cortisol will be measured using Salivette (Sarstedt) devices and analyzed via Chromatography/Mass Spectrometry (nmol/L). Prenatal stress will be assessed using the PES-brief, which consists of two factors measuring distinct positive and negative aspects of pregnancy stress, each each item rated from 0 (not at all) to 3(a great deal). Scoring yields six scores. These are: the frequency of hassles and the frequency of uplifts, intensity of hassles and the intensity of uplifts and two ratio scores Hassles/Uplifts frequencies and Hassles/Uplifts Intensities. Statistical analyses will assess correlations between cortisol levels and PES scores using Pearson's or Spearman's correlation coefficients, while regression models will adjust for confounders.
Correlation Between Neurotrophin Levels and Infant Behavior across study groups | Neurotrophin levels: Maternal serum (15-20 and 36-37 weeks gestation), Umbilical cord blood (at birth) Infant behavior: 6 months postpartum
  This outcome measure examines the correlation between neurotrophin levels (BDNF, Reelin) and infant behavior at 6 months postpartum across the three study groups. Neurotrophin levels will be measured in maternal serum and in umbilical cord blood , using ELISA (pg/mL). Infant behavior will be assessed using the Infant Behavior Questionnaire-Revised Short Form (IBQ-R SF). Statistical analyses will include Spearman's or Pearson's correlation coefficients, with regression models adjusting for confounders.
Correlation Between Neurotrophin Levels and Neonatal Behavior across the study groups | Neurotrophin levels: Maternal serum (15-20 and 36-37 weeks gestation), Umbilical cord blood (at birth) Neonatal behavior: First week of life
  Neurotrophin levels will be measured in maternal serum and in umbilical cord blood , using ELISA (pg/mL. Neonatal behavior will be assessed using the Neonatal Behavioral Assessment Scale (NBAS) during the first week of life. Correlations between neurotrophin levels and NBAS scores will be analyzed using Pearson's or Spearman's correlation coefficients, while regression models will adjust for confounders.Unit of Measure: Neurotrophin levels: pg/mL (ELISA method) Neonatal behavior: NBAS scores
Correlation Between Mother-Child Attachment and Infant Behavior | MPAS assessment: 6 months postpartum IBQ-R SF assessment: 6 months postpartum
  Maternal attachment will be assessed using the Maternal Postnatal Attachment Scale (MPAS), while infant behavior will be evaluated using the Infant Behavior Questionnaire-Revised Short Form (IBQ-R SF). The MPAS consists of 19 items each one ranging from 1 to 5, divided in three constellations : pleasure in interaction, Absence of hostility and Quality of attachment. maximum total score of the scale is 95. Statistical analyses will assess correlations between MPAS and IBQ-R SF scores using Spearman's or Pearson's correlation coefficients, while regression models will adjust for confounders. Unit of Measure: for MPAS score is the sum of the three factors . and for IBQ-R SF score is the Mean score per subscale (temperament domains)

CONTACTS AND LOCATIONS:
Overall Officials: Tania Siahanidou Associate Professor in Pediatrics - Neonatology, MD, PhD, Study Director — 1st_Dept.of Pediatrics_Athens_University_Medical School_Aghia Sophia_Children's Hosp_Athens_11527_GR; Aikaterini Fotiou, MD, MSc, Principal Investigator — Neonatal Dept_Maternity Hosp_Elena Venizelou_2_Plateia Elenas Venizelou Str_Athens 115 21_GR; George P. Chrousos Prof. Emeritus of Pediatrics & Endocrinology_Academician, MD, MACP, MACE, Study Chair — National & Kapodistrian Univ. of Athens_Research_Inst. for Mother-Child Health_Aghia Sophia_Hosp.
Locations (1):
- Maternity Hospital "ELENA VENIZELOU", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected during this study will not be shared with other researchers outside the study team. The data will be used exclusively for statistical analysis by the designated statistician. Data access will remain restricted until the completion, approval, and first official publication of the doctoral dissertation at the university.

REFERENCES:
- [Background] Liang IJ. The wonders of mind-body practices during pregnancy: A topical review. Taiwan J Obstet Gynecol. 2024 Jul;63(4):486-491. doi: 10.1016/j.tjog.2024.04.007. PMID 39004474
- [Background] Alshammari M, Lee RLT, Stubbs M, Chan SW. Effectiveness of psychoeducation interventions for pregnant women with gestational diabetes mellitus: an integrative review. BMC Public Health. 2024 Oct 22;24(1):2929. doi: 10.1186/s12889-024-20428-6. PMID 39438847
- [Background] D'Angelo A, Ceccanti M, Petrella C, Greco A, Tirassa P, Rosso P, Ralli M, Ferraguti G, Fiore M, Messina MP. Role of neurotrophins in pregnancy, delivery and postpartum. Eur J Obstet Gynecol Reprod Biol. 2020 Apr;247:32-41. doi: 10.1016/j.ejogrb.2020.01.046. Epub 2020 Jan 30. PMID 32058187
- [Background] Ardalan M, Chumak T, Quist A, Hermans E, Hoseinpoor Rafati A, Gravina G, Jabbari Shiadeh SM, Svedin P, Alabaf S, Hansen B, Wegener G, Westberg L, Mallard C. Reelin cells and sex-dependent synaptopathology in autism following postnatal immune activation. Br J Pharmacol. 2022 Sep;179(17):4400-4422. doi: 10.1111/bph.15859. Epub 2022 May 23. PMID 35474185
- [Background] Fotiou C, Siahanidou T, Vlastarakos PV, Tavoulari EF, Chrousos G. The effect of body and mind stress-releasing techniques on the breastfeeding of full-term babies; a critical analysis of published interventional studies. J Matern Fetal Neonatal Med. 2018 Jan;31(1):98-105. doi: 10.1080/14767058.2016.1275547. Epub 2017 May 9. PMID 28043180
- [Background] Fotiou C, Vlastarakos PV, Bakoula C, Papagaroufalis K, Bakoyannis G, Darviri C, Chrousos G. Parental stress management using relaxation techniques in a neonatal intensive care unit: A randomised controlled trial. Intensive Crit Care Nurs. 2016 Feb;32:20-8. doi: 10.1016/j.iccn.2015.08.006. PMID 26520208
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Palacios-Garcia I, Lara-Vasquez A, Montiel JF, Diaz-Veliz GF, Sepulveda H, Utreras E, Montecino M, Gonzalez-Billault C, Aboitiz F. Prenatal stress down-regulates Reelin expression by methylation of its promoter and induces adult behavioral impairments in rats. PLoS One. 2015 Feb 13;10(2):e0117680. doi: 10.1371/journal.pone.0117680. eCollection 2015. PMID 25679528
- [Background] Hirota Y, Nakajima K. Control of Neuronal Migration and Aggregation by Reelin Signaling in the Developing Cerebral Cortex. Front Cell Dev Biol. 2017 Apr 26;5:40. doi: 10.3389/fcell.2017.00040. eCollection 2017. PMID 28507985
- [Background] Ranaivoson FM, von Daake S, Comoletti D. Structural Insights into Reelin Function: Present and Future. Front Cell Neurosci. 2016 May 27;10:137. doi: 10.3389/fncel.2016.00137. eCollection 2016. PMID 27303268
- [Background] Boersma GJ, Lee RS, Cordner ZA, Ewald ER, Purcell RH, Moghadam AA, Tamashiro KL. Prenatal stress decreases Bdnf expression and increases methylation of Bdnf exon IV in rats. Epigenetics. 2014 Mar;9(3):437-47. doi: 10.4161/epi.27558. Epub 2013 Dec 23. PMID 24365909
- [Background] Taliaz D, Stall N, Dar DE, Zangen A. Knockdown of brain-derived neurotrophic factor in specific brain sites precipitates behaviors associated with depression and reduces neurogenesis. Mol Psychiatry. 2010 Jan;15(1):80-92. doi: 10.1038/mp.2009.67. Epub 2009 Jul 21. PMID 19621014
- [Background] Malamitsi-Puchner A, Economou E, Rigopoulou O, Boutsikou T. Perinatal changes of brain-derived neurotrophic factor in pre- and fullterm neonates. Early Hum Dev. 2004 Jan;76(1):17-22. doi: 10.1016/j.earlhumdev.2003.10.002. PMID 14729159
- [Background] Claes S. Neuroepigenetics of Prenatal Psychological Stress. Prog Mol Biol Transl Sci. 2018;158:83-104. doi: 10.1016/bs.pmbts.2018.04.007. Epub 2018 Jun 6. PMID 30072061
- [Background] Daskalakis NP, De Kloet ER, Yehuda R, Malaspina D, Kranz TM. Early Life Stress Effects on Glucocorticoid-BDNF Interplay in the Hippocampus. Front Mol Neurosci. 2015 Nov 16;8:68. doi: 10.3389/fnmol.2015.00068. eCollection 2015. PMID 26635521
- [Background] Guan SZ, Fu YJ, Zhao F, Liu HY, Chen XH, Qi FQ, Liu ZH, Ng TB. The mechanism of enriched environment repairing the learning and memory impairment in offspring of prenatal stress by regulating the expression of activity-regulated cytoskeletal-associated and insulin-like growth factor-2 in hippocampus. Environ Health Prev Med. 2021 Jan 15;26(1):8. doi: 10.1186/s12199-020-00929-7. PMID 33451279
- [Background] Guan SZ, Ning L, Tao N, Lian YL, Liu JW, Ng TB. Effects of maternal stress during pregnancy on learning and memory via hippocampal BDNF, Arc (Arg3.1) expression in offspring. Environ Toxicol Pharmacol. 2016 Sep;46:158-167. doi: 10.1016/j.etap.2016.04.012. Epub 2016 Jun 29. PMID 27474832
- [Background] Conradt E, Adkins DE, Crowell SE, Raby KL, Diamond LM, Ellis B. Incorporating epigenetic mechanisms to advance fetal programming theories. Dev Psychopathol. 2018 Aug;30(3):807-824. doi: 10.1017/S0954579418000469. PMID 30068415
- [Background] Sandman CA, Davis EP, Buss C, Glynn LM. Exposure to prenatal psychobiological stress exerts programming influences on the mother and her fetus. Neuroendocrinology. 2012;95(1):7-21. doi: 10.1159/000327017. Epub 2011 Apr 15. PMID 21494029
- [Background] Creutzberg KC, Sanson A, Viola TW, Marchisella F, Begni V, Grassi-Oliveira R, Riva MA. Long-lasting effects of prenatal stress on HPA axis and inflammation: A systematic review and multilevel meta-analysis in rodent studies. Neurosci Biobehav Rev. 2021 Aug;127:270-283. doi: 10.1016/j.neubiorev.2021.04.032. Epub 2021 May 2. PMID 33951412
- [Background] Grundwald NJ, Brunton PJ. Prenatal stress programs neuroendocrine stress responses and affective behaviors in second generation rats in a sex-dependent manner. Psychoneuroendocrinology. 2015 Dec;62:204-16. doi: 10.1016/j.psyneuen.2015.08.010. Epub 2015 Aug 17. PMID 26318631
- [Background] Hernandez-Reif M, Kendrick A, Avery DM. Pregnant women with depressive and anxiety symptoms read, talk, and sing less to their fetuses. J Affect Disord. 2018 Mar 15;229:532-537. doi: 10.1016/j.jad.2017.12.108. Epub 2018 Jan 5. No abstract available. PMID 29353212
- [Background] Vega-Sanz M, Rey-Saez R, Berastegui A, Sanchez-Lopez A. Difficulties in Pregnancy Adjustment as Predictors of Perinatal Depression: Indirect Effects through the Role of Brooding Rumination and Maternal-Fetal Bonding. Am J Perinatol. 2024 May;41(S 01):e2870-e2877. doi: 10.1055/s-0043-1776062. Epub 2023 Oct 17. PMID 37848044
- [Background] Witt WP, Litzelman K, Cheng ER, Wakeel F, Barker ES. Measuring stress before and during pregnancy: a review of population-based studies of obstetric outcomes. Matern Child Health J. 2014 Jan;18(1):52-63. doi: 10.1007/s10995-013-1233-x. PMID 23447085
- [Background] Lau C. Effects of stress on lactation. Pediatr Clin North Am. 2001 Feb;48(1):221-34. doi: 10.1016/s0031-3955(05)70296-0. No abstract available. PMID 11236728
- [Background] Tavoulari EF, Benetou V, Vlastarakos PV, Psaltopoulou T, Chrousos G, Kreatsas G, Gryparis A, Linos A. Factors affecting breastfeeding duration in Greece: What is important? World J Clin Pediatr. 2016 Aug 8;5(3):349-57. doi: 10.5409/wjcp.v5.i3.349. eCollection 2016 Aug 8. PMID 27610353
- [Background] Atchan M, Davis D, Foureur M. The impact of the Baby Friendly Health Initiative in the Australian health care system: a critical narrative review of the evidence. Breastfeed Rev. 2013 Jul;21(2):15-22. PMID 23957177
- [Background] Skouteris H, Bailey C, Nagle C, Hauck Y, Bruce L, Morris H. Interventions Designed to Promote Exclusive Breastfeeding in High-Income Countries: A Systematic Review Update. Breastfeed Med. 2017 Dec;12(10):604-614. doi: 10.1089/bfm.2017.0065. Epub 2017 Sep 8. PMID 28885859
- [Background] Bartick MC, Schwarz EB, Green BD, Jegier BJ, Reinhold AG, Colaizy TT, Bogen DL, Schaefer AJ, Stuebe AM. Suboptimal breastfeeding in the United States: Maternal and pediatric health outcomes and costs. Matern Child Nutr. 2017 Jan;13(1):e12366. doi: 10.1111/mcn.12366. Epub 2016 Sep 19. PMID 27647492
- [Background] Mimouni FB, Koletzko B. Human Milk for Preterm Infants. Clin Perinatol. 2017 Mar;44(1):xix-xx. doi: 10.1016/j.clp.2016.12.001. No abstract available. PMID 28159213
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- Available data/document: Peer-reviewed journal publication related to the study: 10.47363/JPRRR/2024(6)163 — https://onlinescientificresearch.com/articles/greek-validation-of-the-questionnaire-prenatal-breastfeeding-self-efficacy-scale.pdf — Greek Validation of the Questionnaire "Prenatal Breast-Feeding Self Efficacy" Scale July 2024Journal of Pediatrics Research Reviews & Reports
- Available data/document: Peer-reviewed journal publication related to the study: PMID: 28043180 — https://pubmed.ncbi.nlm.nih.gov/28043180/ — Title: The effect of body and mind stress-releasing techniques on the breastfeeding of full term babies; a critical analysis of published interventional studies